CLINICAL TRIAL: NCT05367895
Title: Effectiveness of CoronaVac® First Booster Dose for Preventing Symptomatic Acute Respiratory Infection Caused by SARS-CoV-2 Virus in Adults in São Paulo City, Brazil: a Retrospective Test-negative Case-control Study
Brief Title: Effectiveness of Inactivated COVID-19 Vaccine of the First Booster Dose
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Other Study IDs: EFFERVESCENCE/ BRAZIL
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The samples without DNA. Only data will be recovered from three health surveillance information electronic health records:
  1. VACIVIDA, comprising individual data for people vaccinated against SARS-Cov-2.
  2. E-SUS, mandatory report database for mild to moderate COVID-19.
  3. SIVEP-GRIPE, mandatory report database for severe cases of COVID-19 All those RWD sources are available at the São Paulo Municipality Centers for Health Surveillance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Exposure group 1: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022 and received a three-dose homologous vaccination with CoronaVac. Specifically, ≥14 days after receipt of the third vaccine dose using a homologous regimen with CoronaVac.
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- Exposure group 2: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who received a two-dose vaccination with CoronaVac and did not receive any booster vaccine. Specifically, ≥14 days after receipt of the second vaccine dose and before the third dose of CoronaVac.
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- Exposure group 3: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who received only one dose vaccination with CoronaVac and did not receive any other vaccine dose. Specifically, ≥14 days after receipt of the first vaccine dose and before the second dose of CoronaVac.
- Non-Exposure group: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who were not vaccinated. No history of vaccination for any type of COVID-19 vaccine, or <14 days after receipt of the first vaccine of CoronaVac.
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — Form: CoronaVac® is a milky-white suspension. Stratified precipitate may form that can be dispersed by shaking.
  Presentation: Each vial contains 0.5 mL (a single dose) and contains 600SU of inactivated SARS-CoV-2 virus antigen.
  Administration and schedule: Two doses with an interval of 21 days should be administered for primary immunization. 0.5 mL per dose.
  Route: IM in the deltoid region of the upper arm after shaking the vial well before use.
  Other Names: CoronaVac®
  Groups: Exposure group 1; Exposure group 2; Non-Exposure group

SUMMARY:
This is a retrospective test-negative case-control study of COVID-19 Vaccine (CoronaVac®) manufactured by Sinovac Research and Development Co., Ltd.The main purpose of this study is to measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed symptomatic disease.

DETAILED DESCRIPTION:
This is a retrospective test-negative case-control study in São Paulo city, Brazil . The COVID-19 Vaccine (CoronaVac® )produced by Sinovac Research and Development Co., Ltd.The main purpose of this study is to measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed symptomatic disease.A total of 14000 subjects will be enrolled,including 7,000 positive cases and 7,000 test negative COVID-19 cases The Statistical Analysis Plan (SAP) will include univariate (and, when required, multivariable) models of logistic regression.Data will be recovered from three health surveillance information electronic health records (EHRs):

1. VACIVIDA, comprising individual data for people vaccinated against SARS-Cov-2.
2. E-SUS, mandatory report database for mild to moderate COVID-19.
3. SIVEP-GRIPE, mandatory report database for severe cases of COVID-19. All those RWD sources are available at the São Paulo Municipality Centers for Health Surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Exposure group 1: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022 and received a three-dose homologous vaccination with CoronaVac. Specifically, ≥14 days after receipt of the third vaccine dose using a homologous regimen with CoronaVac.
* Exposure group 2: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who received a two-dose vaccination with CoronaVac and did not receive any booster vaccine. Specifically, ≥14 days after receipt of the second vaccine dose and before the third dose of CoronaVac.
* Exposure group 3: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who received only one dose vaccination with CoronaVac and did not receive any other vaccine dose. Specifically, ≥14 days after receipt of the first vaccine dose and before the second dose of CoronaVac.
* Non-Exposure group: Adults (≥ 18 years of age) registered in the E-SUS or SIVEP-gripe RWD source data from August 16th, 2021 through April 21st, 2022, who were not vaccinated. No history of vaccination for any type of COVID-19 vaccine, or <14 days after receipt of the first vaccine of CoronaVac.

Exclusion Criteria:

* Anyone who received other vaccines for the first doses.
* Anyone who received CoronaVac for the two initial doses but other vaccines for the booster (heterologous immunization).
* Subjects with incomplete vaccination history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is community-dwelling individuals aged 18 years and above with no contra-indication for COVID-19 vaccination who consult a participating general practitioner or a hospital in São Paulo city, Brazil if they develop illness of interests (i.e., WHO definition of suspected COVID-19 cases) and had RT-PCR for SARS-Cov-2 colleceted.
Sampling Method: Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of homologous booster-dose vaccination with CoronaVac® | 6 months after the third dose of COVID-19 vaccine
  To measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed symptomatic disease

SECONDARY OUTCOMES:
effectiveness of homologous booster-dose vaccination with CoronaVac® | 6 months after the third dose of COVID-19 vaccine
  To measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed COVID-19 hospital admissions
vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® | 6 months after the third dose of COVID-19 vaccine
  To measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed COVID-19 intensive care unit admissions.
Vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® | 6 months after the third dose of COVID-19 vaccine
  To measure vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® against laboratory-confirmed COVID-19 intensive care unit deaths.

OTHER OUTCOMES:
vaccine effectiveness of homologous booster-dose vaccination | 6 months after the third dose of COVID-19 vaccine
  To compare vaccine effectiveness of homologous booster-dose vaccination with CoronaVac® in periods with predominance of Delta and Omicron SARS-CoV-2 variants
help support the approval of new indication (i.e. boosters) of the CoronaVac®. | 6 months after the third dose of COVID-19 vaccine
  To generate data to help support the approval of new indication (i.e. boosters) of the CoronaVac®.
support post-approval study requirements of CoronaVac®. | 6 months after the third dose of COVID-19 vaccine
  To support post-approval study requirements of CoronaVac®.

CONTACTS AND LOCATIONS:
Overall Officials: André Machado amsiqueira@gmail.com, Doctor, Principal Investigator — amsiqueira@gmail.com
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas (INI-FIOCRUZ), Manguinhos, Brazil